CLINICAL TRIAL: NCT07372677
Title: Clinical and Microbiological Effects of a Thermal-Gel Device in Periodontal Treatment: Diabetic vs Non-Diabetic Patients
Brief Title: Pocket-X Gel Non-surgical Periodontal Therapy
Acronym: DEFECT_PERIO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Collaborators: University of Verona, Italy (Unknown)
Responsible Party: Principal Investigator, Alessia Pardo, PhD, Universita di Verona
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 590CET; Etics Commitee (Registry Identifier: Etics Commitee for Clinical Trials of the Provinces Verona and Rovigo)
Record Dates: First submitted 2026-01-19; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Diabete Type 2
Keywords: Non-surgical periodontal therapy; Pocket-X gel; Periodontits in diabete type-2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The study is clinical, with the following characteristics: prospective, case-control, single-center, with a post-market device. The case group is represented by patients affected by controlled T2DM, the control group by non-diabetic patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gel therapy after non surgical therapy (Experimental): The test group will receive gel therapy immediately after non surgical treatment. The gel in use is a composition of Hyaluronic acid, Poloxamer, 2-Phenoxyethanol, Octedine HCL,Water (Pocket-X Gel Geistlich AG, Wolhusen, Switzerland). It is a patented liquid-to-gel device. Pocket-X® Gel is composed of: Poloxamer 407 with thermo-gelling properties, Octenidine, antimicrobial preservative, Hyaluronic acid to support tissue healing.
  Interventions: Device: Gel therapy after non surgical therapy
- Non surgical therapy (No Intervention): In the control group non surgical therapy was performed using mechanical and manual instrumentations (curettes and ultrasonic devices)

INTERVENTIONS:
Device: Gel therapy after non surgical therapy — The gel in use is a composition of Hyaluronic acid, Poloxamer, 2-Phenoxyethanol, Octedine HCL,Water (Pocket-X Gel Geistlich AG, Wolhusen, Switzerland). It is a patented liquid-to-gel device. Pocket-X® Gel is composed of: Poloxamer 407 with thermo-gelling properties, Octenidine, antimicrobial preservative, Hyaluronic acid to support tissue healing. It promotes gingival healing and prevents bacterial recolonization of periodontal pockets, forming a protective physical barrier, allows to postpone or avoid long, complex and painful surgeries, ensuring the success of periodontal treatment, delaying any surgical interventions.
  Arms: Gel therapy after non surgical therapy

SUMMARY:
Evaluate from a clinical and microbiological point of view the effect of an adjunctive therapy based on a thermal-gelling device Pocket-X® Gel (Hyaluronic acid, Poloxamer, 2-Phenoxyethanol, Octedine HCL, Water), in the non-surgical treatment of periodontal defects, in a population of patients with T2DM compared to non-diabetic patients.

Determine whether periodontal defect healing is clinically and microbiologically different between T2DM patients and non-diabetic patients; whether periodontal treatment and maintenance can lead to improvement of conditions and stability over time also for diabetic conditions.

ELIGIBILITY:
Inclusion Criteria:

Patients normally eligible for the visit and for the non-surgical type of treatment for periodontal defects:

* patients with an age between 18 and 80;
* patients with: (i) Asa status I (no functional impairment due to pathologies), (ii) patients with type 2 diabetes (T2DM) with: glycated hemoglobin level HbA1c between 6.5 and 8.0%, on dietary therapy and/or with hypoglycemic drugs in regular follow-up at the diabetes service;
* patients with chronic periodontitis stage 3 or 4, according to the new classification of periodontal diseases [Tonetti et al.]), verified clinically and radiographically: patients will be selected with interdental clinical attachment level (CAL) at the site of greatest loss ≥3 mm to ≥2 non-adjacent teeth, probing depth (PPD) ≥5 mm, bleeding on probing (BoP) and horizontal and/or vertical radiographic bone loss.

Exclusion Criteria:

* Patients not eligible for the non-surgical type of treatment for periodontal defects:

  * patients with a positive history of diseases with functional impairment (ASA status 2,3,4) or severe handicaps that could limit the ability to attend appointments;
  * patients with uncontrolled/poorly controlled DM at the time of study selection (e.g. type 1 diabetes mellitus and secondary forms of diabetes); patients with uncontrolled and serious diabetic complications (cardiovascular, renal, hepatic and nervous);
  * poor compliance with treatment, with poor oral hygiene and motivation;
  * not signing informed consent by patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation, in the test site and in the control site (for each of the two groups) of the periodontal index of: PPD in mm. | At baseline and after 2 weeks, 1 month, and 3 months
  Clinical evaluation, in the test site and in the control site (for each of the two groups), at baseline and after 2 weeks, 1 month, and 3 months, by means of detection with a periodontal millimeter probe, of the periodontal index of: pocket probing depth (PPD), in mm.
  Detect whether the healing of periodontal defects is different from a clinical and microbiological point of view between patients with T2DM and non-diabetic patients; whether periodontal treatment and maintenance can bring improvement of conditions and stability over time also for the diabetic condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Alessia Pardo 3494628471 Alessia.pardo@univr.it, Verona, Italy, Italy